CLINICAL TRIAL: NCT01412216
Title: The Effects of Sedentarism on Vascular Function, Inflammation, and Insulin Resistance
Acronym: Bedrest
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding Depleted.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Sedentarism
Record Dates: First submitted 2011-08-05; First posted 2011-08-09 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Endothelial Dysfunction; Insulin Resistance; Metabolic Syndrome; Peripheral Arterial Disease
Keywords: Sedentarism; Physical inactivity; Fish oil; Omega-3 fatty acids; Endothelial dysfunction; Insulin resistance; Metabolic syndrome; peripheral arterial disease
MeSH Terms: conditions — Insulin Resistance; Metabolic Syndrome; Peripheral Arterial Disease; Sedentary Behavior | interventions — Fish Oils; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Fish Oil (Omega-3 Fatty Acids) (Experimental): High-dose, short-duration dietary omega-3 fatty acids supplementation
  Interventions: Dietary Supplement: Fish Oil (Omega-3 Fatty Acids)
- Placebo (Placebo Comparator): Placebo control
  Interventions: Dietary Supplement: Fish Oil (Omega-3 Fatty Acids)

INTERVENTIONS:
Dietary Supplement: Fish Oil (Omega-3 Fatty Acids) — fish oil-4.4gm/day x 5 days
  Arms: Fish Oil (Omega-3 Fatty Acids)
Dietary Supplement: Fish Oil (Omega-3 Fatty Acids)
  Arms: Placebo

SUMMARY:
The purpose of this study are twofold:

1. To understand the effects of physical inactivity (sedentarism) on vascular function, insulin resistance and inflammation;
2. To assess the role of a dietary intervention (fish oil) in counteracting the effects of physical inactivity on vascular function and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects: Subjects must be free from any acute, chronic or debilitating medical conditions. Healthy status will be established on the basis of clinical history, electrocardiogram, clinical biochemical screening tests of blood and urine, a physical examination, and where necessary a chest radiograph.

Exclusion Criteria:

* Any active acute or chronic medical problem: Any subject with symptoms of active illness (e.g., fever, leukocytosis, hypertension) will be excluded from study. The exclusion criteria will also include history or evidence for psychiatric disorders, hypertension, diabetes, coronary artery disease (CAD), renal insufficiency, thyroid disease, alcohol or drug abuse, viral hepatitis, deep venous thrombosis or anemia. Individuals with a history of psychiatric illnesses or psychiatric disorders will also be excluded, such as alcoholism, drug dependency including dependency on tobacco, major mood disorders such as major depression and manic depressive illness, schizophrenic disorders, anxiety disorders including panic disorder, generalized anxiety disorder, post traumatic stress disorder, obsessive compulsive disorder, agoraphobia, claustrophobia, paranoid personality disorder, schizoid personality disorder, schizotypal personality disorder, borderline personality disorder, and antisocial personality disorder. In addition, potential subjects with a first order relative with a history of major depressive illness, manic depressive illness, schizophrenia, agoraphobia or panic disorder will also be excluded from entry to this study. Finally, individuals who are unaware of specific psychiatric diagnoses who have a history of having been treated with antidepressant, neuroleptic medications or major tranquilizers will be excluded from study. However, a personal history of limited prior counseling or psychotherapy (e.g., for adjustment reactions) will not necessarily be exclusionary.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2011-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Endothelial Function | 5 days
  Flow-mediated, brachial artery vasodilation (FMD)

SECONDARY OUTCOMES:
Insulin Resistance | 5 days
  The homeostatic model assessment (HOMA) method used to quantify insulin resistance (HOMA-IR)

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Grenon, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States